CLINICAL TRIAL: NCT03629964
Title: Real-Time Head Position Stabilization of Patients Undergoing Radiation Therapy
Brief Title: Study to Develop Head Stabilizer for Use During Brain Radiation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left site.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB17-0506
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Brain Diseases; Brain Cancer
MeSH Terms: conditions — Brain Diseases; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Head stabilizer group (Experimental): Patients will be receiving standard brain radiation. The experimental head holder device (called the Wiersma Head Stabilizer) will be attached to treatment table and will make small movements to adjust the position of the head in response to movement by the patient. In addition, the AlignRT system (an FDA approved medical device that automatically turns off the radiation beam if the patient's head moves beyond a set distance) will be used to track real-time motions of the head. This system is used with radiation therapy as standard of care.
  Interventions: Device: Wiersma Head Stabilizer; Device: AlignRT system

INTERVENTIONS:
Device: Wiersma Head Stabilizer — Experimental device attached to treatment table.
Device: AlignRT system — The AlignRT system (an FDA approved medical device that automatically turns off the radiation beam if the head moves beyond a set distance) will be used to track real-time motions of the head. This system is used with radiation therapy as standard of care.

SUMMARY:
The purpose of this study is to begin to develop a device to stabilize the head during stereotactic radiosurgery (SRS). SRS is a therapy for brain disorders and cancers that uses a precise dose of radiation to treat a disease, and is different from whole brain radiation. This study aims to stabilize patient head motions during radiation therapy through the use of a special experimental head holder. The investigators would like to first see how the experimental device works in whole brain radiation.

ELIGIBILITY:
Adults undergoing whole brain radiation cancer treatment at the University of Chicago Medicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Access feasibility of the use of an experimental head stabilizer device | During radiation treatment (5-10 days)
  Feasibility will be defined as to whether or not the 6D target is ≤ 0.5mm and ≤ 0.5deg for greater than 95% of treatment time

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Wiersma, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided